CLINICAL TRIAL: NCT04304443
Title: Non Traumatic Aortic Dissection : Chain of Care and Pre-hospital Risk Factors, a Retrospective, Multicenter Study
Brief Title: Pre-hospital Management of Aortic Dissection
Acronym: FFDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Hopital Nord Franche-Comte (Other); Centre Hospitalier de Lons Le Saunier (Unknown); Centre hospitalier de Vesoul (Unknown); Centre hospitalier de Pontarlier (Unknown); Centre hospitalier de Gray (Unknown); Centre hospitalier de Dole (Unknown); Centre Hospitalier de Saint-Claude (Unknown)
Responsible Party: Sponsor
Other Study IDs: P/2019/453
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-02

CONDITIONS: Aortic Dissection
Keywords: Aortic Dissection; Mortality; Treatment delay; Emergency; Pre-hospital phase
MeSH Terms: conditions — Aortic Dissection; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background :

Time between symptoms onset and treatment initiation is crucial in Acute aortic dissection (AAD). An anti-hypertensive treatment can be rapidly initiated before the arrival in Emergency Department (ED). A better understanding of the chain of care between symptoms onset and surgery could lead to a reduction of morbi-mortality. Our study have the objective to describe the chain of care of patients with AAD in the ED.

Methods :

This is an observational, retrospective, multicenter study. Patients were detected with a discharge of diagnostic of aortic dissection (ICD I71.0) in university medical center of Besançon. Data collection : patients records in the 8 hospitals centers of the area Franche-Comté.

DETAILED DESCRIPTION:
Acute aortic dissection (AAD) is the most lethal vascular emergency. AAD remains a challenge to diagnose and to treat even for experienced practitioners. AAD identification and treatment administration greatly improve morbidity and mortality associated to AAD. The diagnosis of AAD is particularly challenging, due to a combination of highly heterogeneous clinical presentation and low incidence (3-5 cases/100,000 individuals/year). Clinical guidelines suggest that AAD should be considered in all patients presenting with chest pain, back pain, abdominal pain, syncope or symptoms consistent with perfusion deficit, but these symptoms account for large proportions of emergency medical visits. CT-scan is validated and increasedly available for confirming or ruling out AAD. Stanford classification is most current use, with two groups : type A involve the ascending aorta, type B don't involve the ascending aorta until the arch. The majority of type A is managed surgically, but the majority of type B is managed medically with anti-hypertensive treatment. Aortic dissection can be classified into hyperacute (from symptom onset to 24 hours), acute (2-7 days), subacute (8-30 days), and chronic (> 30 days). Booher et al, suggested that acute and sub-acute aortic dissection make the majority of the mortality rate.

Mortality among patients with a Stanfond Type A dissection is 1 to 2 percent per hour, early after symptom onset. In-hospital mortality is highly dependent on patient risk profiles before surgery. Patient with a history of aortic valve replacement, a migrating chest pain, a tamponade, an hypotension or a limb ischemia are associated to a higher in-hospital mortality.

Time between symptoms onset and treatment initiation is crucial. The diagnosis can be suspected by the family physician. In France, diagnosis can be also suspected by the MICU (Mobile Intensive Care Unit). An anti-hypertensive treatment can be rapidly initiated before the arrival by the ED, and the diagnosis is confirmed by CT-scan. In the Harris' study, median time from arrival at the emergency department to diagnosis and from diagnosis to surgery were 4.3 hours. To our knowledge no study investigated the pre-hospital phase, especially the impact of the methods and vectors used. A better understanding of the chain of care from symptoms onset to surgery could lead to a reduction of morbi-mortality. Our study aimed the objective to describe the chain of care of patients with AAD in the ED of eight hospitals centers of area of Franche-Comté (France) between 2010 and 2019.

ELIGIBILITY:
Inclusion Criteria :

* patients with age > 18 years
* patients with the diagnosis of non traumatic acute aortic dissection
* patients hospitalized in the university medical center

Exclusion Criteria :

* decision of withdrawal life support
* patients that died without a diagnosis confirmation with Helical Computed Tomography (HCT), Magnetic Resonnance Imagery (MRI), TransEsophageal Echocardiography (TEE) or surgery/autopsy
* AAD that were complications of coronarography or aortic surgery
* lack of information
* patient opposition to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients supported for an AAD between 2010-2019 in one of height hospitals centers participants.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Daguerre, MD-student, Principal Investigator — CHU de Besançon; Antoine Sigaux, MD, Study Director — CHU de Besançon; Thibaut Desmettre, MD, PHD, Study Chair — CHU de Besançon
Locations (2):
- France (2):
  - CHU de Besançon, Besançon
  - Hôpital Nord Franche-Comté, Trévenans

REFERENCES:
- [Result] Axelsson C, Karlsson T, Pande K, Wigertz K, Ortenwall P, Nordanstig J, Herlitz J. A description of the prehospital phase of aortic dissection in terms of early suspicion and treatment. Prehosp Disaster Med. 2015 Apr;30(2):155-62. doi: 10.1017/S1049023X15000060. Epub 2015 Feb 10. PMID 25668482
- [Result] Dixon M. Misdiagnosing aortic dissection: a fatal mistake. J Vasc Nurs. 2011 Dec;29(4):139-46. doi: 10.1016/j.jvn.2011.08.003. PMID 22062792
- [Result] Nazerian P, Giachino F, Vanni S, Veglio MG, Castelli M, Lison D, Bitossi L, Moiraghi C, Grifoni S, Morello F. Diagnostic performance of the aortic dissection detection risk score in patients with suspected acute aortic dissection. Eur Heart J Acute Cardiovasc Care. 2014 Dec;3(4):373-81. doi: 10.1177/2048872614527010. Epub 2014 Mar 6. PMID 24604712
- [Result] Pape LA, Awais M, Woznicki EM, Suzuki T, Trimarchi S, Evangelista A, Myrmel T, Larsen M, Harris KM, Greason K, Di Eusanio M, Bossone E, Montgomery DG, Eagle KA, Nienaber CA, Isselbacher EM, O'Gara P. Presentation, Diagnosis, and Outcomes of Acute Aortic Dissection: 17-Year Trends From the International Registry of Acute Aortic Dissection. J Am Coll Cardiol. 2015 Jul 28;66(4):350-8. doi: 10.1016/j.jacc.2015.05.029. PMID 26205591
- [Result] Harris KM, Strauss CE, Eagle KA, Hirsch AT, Isselbacher EM, Tsai TT, Shiran H, Fattori R, Evangelista A, Cooper JV, Montgomery DG, Froehlich JB, Nienaber CA; International Registry of Acute Aortic Dissection (IRAD) Investigators. Correlates of delayed recognition and treatment of acute type A aortic dissection: the International Registry of Acute Aortic Dissection (IRAD). Circulation. 2011 Nov 1;124(18):1911-8. doi: 10.1161/CIRCULATIONAHA.110.006320. Epub 2011 Oct 3. PMID 21969019
- [Result] Evangelista A, Isselbacher EM, Bossone E, Gleason TG, Eusanio MD, Sechtem U, Ehrlich MP, Trimarchi S, Braverman AC, Myrmel T, Harris KM, Hutchinson S, O'Gara P, Suzuki T, Nienaber CA, Eagle KA; IRAD Investigators. Insights From the International Registry of Acute Aortic Dissection: A 20-Year Experience of Collaborative Clinical Research. Circulation. 2018 Apr 24;137(17):1846-1860. doi: 10.1161/CIRCULATIONAHA.117.031264. PMID 29685932
- [Result] Booher AM, Isselbacher EM, Nienaber CA, Trimarchi S, Evangelista A, Montgomery DG, Froehlich JB, Ehrlich MP, Oh JK, Januzzi JL, O'Gara P, Sundt TM, Harris KM, Bossone E, Pyeritz RE, Eagle KA; IRAD Investigators. The IRAD classification system for characterizing survival after aortic dissection. Am J Med. 2013 Aug;126(8):730.e19-24. doi: 10.1016/j.amjmed.2013.01.020. PMID 23885677